CLINICAL TRIAL: NCT02164890
Title: Pharmacokinetics of Micafungin in Patients of Intensive Care Units
Acronym: MI-K
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: I13025
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2016-06

CONDITIONS: Invasive Candidiasis
MeSH Terms: conditions — Candidiasis, Invasive | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmacokinetics of micafungin (Other)
  Interventions: Other: micafungin

INTERVENTIONS:
Other: micafungin — This is a pharmacokinetic study where a total number of 14 blood samples will be drawn per patient. Clinical and biological data will be concomitantly collected.

SUMMARY:
Invasive fungal infections (IFIs) are a frequent cause of morbidity and mortality in high-risk patients, such as immunocompromised patients. Candida is currently the predominant fungal pathogen in these patient populations and is associated with significant morbidity and a high mortality.

Micafungin (MCF) is a semisynthetic compound belonging to the new class of antifungal agents, the echinocandin lipopeptides, that has potent in vitro and experimental in vivo activity against a variety of pathogenic Candida species and Aspergillus species. Its applied indications are so the treatment and/or the prophylaxis of Candida and Aspergillus infections. MCF is currently licensed for the treatment of candidiasis at doses of either 100 or 150 mg a day.

The efficacy of MCF is linked to the area under the concentration-time curve over 24 h in the steady state divided by the MIC (AUC0-24/ MIC ratio).

On one hand:

- It was demonstrated that 98% of invasive candidiasis patients with a MCF AUC/MIC ratio between 3 and 12 achieve microbiological clearance, as opposed to only 85% of those with an AUC/MIC ratio < 3. In the case of infections by Candida parapsilosis, which exhibits drug MICs that are 50- to100-fold higher, 100% of patients with an AUC/MIC ratio >285 achieve microbiological clearance, as opposed to 82% of those below that exposure level.(1)

On the other hand:

* It is well known that patients of intensive care units (ICU) are characterized by particular pharmacokinetic parameters with higher apparent volume of distribution (VC/F) and/or higher apparent systemic clearance (CL/F). In a population of healthy volunteers, it was observed that CL/F of MCF presents a high interpatient variability.(2)
* Whether most ICUs patients achieve optimal AUC/MIC ratio thresholds at standard doses has not been investigated so far. In particular, lower AUCs might be reached in patients having the highest VC/F values. Such patients would then be at risk of therapy failure and would benefit from individualized-dosing strategies.

In this context, the study of the pharmacokinetics of MCF in critically ill patients seems to be necessary.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients hospitalized in an ICU, with suspected or proven invasive fungal infections, for whom the decision has been made to start a treatment based on MCF.
* Age > 18 years.
* Patients willing to give their written informed consent for their participation to the study.
* Patients affiliated to the French social security system or equivalent.

Exclusion Criteria:

* Patient for whom a treatment based on MCF has already been started
* Patient who have benefited from bone marrow transplantation
* Age < 18 years
* Patient under legal protection
* Patient deprived of liberty
* Pregnant or breast-feeding woman or woman of childbearing potential without efficient contraception (based on declaration)
* Patient with any altered mental status or any psychiatric condition that would interfere with the understanding of the study
* Patient enrolled in another clinical trial testing drugs or therapeutic strategies (including the so-called "exclusion period")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To describe micafungin concentrations over time, | 3 weeks
  The evaluation of the PK model performance will be based on its ability:
  * To describe micafungin concentrations over time,
  * To explain the sources of inter-individual PK variability. It will be done by the calculation of the bias between concentrations predicted using the model and observed concentrations.

SECONDARY OUTCOMES:
To estimate the proportion of patients hospitalized in an ICU achieving the target AUC or AUC/MIC when receiving the recommended regimen | 3 weeks
  The estimation of the proportion of patients hospitalized in an ICU achieving the target AUC or AUC/MIC when receiving the recommended regimen will be based on the determination of exposure indices (AUC) and mycological characteristics (fungus and its MIC)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Montpellier, Montpellier, France

REFERENCES:
- [Result] Berrah R, Saint-Marcoux F, Monchaud C, Cointault O, Conseil M, Jaber S, Jung B, Woillard JB. From AUC/MIC to AUCss and Cmin: Optimizing Micafungin Therapy in the Critically Ill through Model-Informed Precision Dosing. AAPS J. 2025 Nov 11;28(1):18. doi: 10.1208/s12248-025-01173-z. PMID 41219680